CLINICAL TRIAL: NCT00248833
Title: Phase 1 Dose Esc Study of Safety and Immun of 3 Injections, Given at 0, 6 and 24 Wks, of Grp B Meningococcal 44/76 MOS NOMV 5D Vaccine Admin to Healthy Subjs IM With and Without Adjuvant
Brief Title: Safety and Immunogenicity Study of Group B Meningococcal Vaccine to Prevent Meningitis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRAIR 1178; HSRRB A-13513
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-01

CONDITIONS: Meningitis, Meningococcal, Serogroup B
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Intervention Model Description: The study was conducted as a phase 1, outpatient, dose-escalating study for the Meningococcal 44/76 MOS NOMV 5D Vaccine (lot number 1119). Two dosage levels were investigated: 25 µg with and without adjuvant and 50 µg of protein without adjuvant. Each dose was given intramuscularly at 0, 6, and 24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The first 2 cohorts were double blind, and the third cohort was not blinded. The investigator preparing the vaccine did not participate in making subsequent study assessments or subject evaluability decisions. After the vaccine was prepared, the subject's identification number was placed onto the drawn syringe. All information, vaccine dose, adjuvant dose (if applicable), and subject identification number, was recorded on the Vaccine Administration Code Form. The form was placed in an envelope. The envelope was sealed and placed in a secured location. The medical personnel who vaccinated the subjects witnessed the dilution and placement of the subject identification number on the syringe. This staff member vaccinated the subject but did not participate in subsequent study visits or the evaluation. The blind was broken after verification that all serology testing was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o adjuvant (Experimental): Subjects received 25ug Group B Meningococcal 44/76 MOS NOMV 5D without AI (OH)3 adjuvant intramuscularly at 0, 6, and 24 weeks.
  Interventions: Biological: 25ug Group B Meningococcal 44/76 MOS NOMV 5D Vaccine
- 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D with adjuvant (Experimental): Subjects received 25ug Group B Meningococcal 44/76 MOS NOMV 5D with AI (OH)3 adjuvant intramuscularly at 0, 6, and 24 weeks.
  Interventions: Biological: 25ug Group B Meningococcal 44/76 MOS NOMV 5D Vaccine
- 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o adjuvant (Experimental): Subjects received 50ug Group B Meningococcal 44/76 MOS NOMV 5D without AI (OH)3 adjuvant intramuscularly at 0, 6, and 24 weeks.
  Interventions: Biological: 50ug Group B Meningococcal 44/76 MOS NOMV 5D Vaccine

INTERVENTIONS:
Biological: 25ug Group B Meningococcal 44/76 MOS NOMV 5D Vaccine — The study was conducted as a phase 1, outpatient, dose-escalating study for the Meningococcal 44/76 MOS NOMV 5D Vaccine (lot number 1119). 25µg with and without adjuvant were administered. Vaccinations were given intramuscularly at 0, 6, and 24 weeks.
  Arms: 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o adjuvant; 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D with adjuvant
Biological: 50ug Group B Meningococcal 44/76 MOS NOMV 5D Vaccine — The study was conducted as a phase 1, outpatient, dose-escalating study for the Meningococcal 44/76 MOS NOMV 5D Vaccine (lot number 1119). 50µg without adjuvant was administered. Vaccinations were given intramuscularly at 0, 6, and 24 weeks.
  Arms: 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o adjuvant

SUMMARY:
The purpose of this study is to determine if the vaccine called Group B Meningococcal 44/76 MOS NOMV 5D Vaccine is safe and free from side effects and if it will protect people from meningitis.

This study will vaccinate three groups of people. In the first 2 groups, the study will be double-blinded. This means that neither the volunteer or the medical team will know which formulation of the vaccine was administered. The third group of volunteers and the medical team will know that they are receiving the higher dose of the vaccine.

DETAILED DESCRIPTION:
Meningococcal disease is a contagious bacterial disease caused by Neisseria meningitidis that can kill children and young adults very quickly. Meningococci are divided into distinct sergroups based on their polysaccharide outer capsule, which is the usual target antigen for vaccines. Serogroup A is the main cause of epidemics in Africa and in the United States, sergroups B, C and Y predominate. In the United States, no vaccine is yet available to offer protection against serogroup B which currently accounts for 32% of all meningococcal disease in the United States.

This study serves as a proof of concept for our new NOMV Group B single strain monovalent vaccine model which is obtained from a genetically modified parent. If successful we plan to develop a multivalent Group B vaccine for routine use for military recruits at the beginning of basic training, for college students, particularly those who live in dormitories, and for use by travelers to countries recognized as having hyperendemic disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy military or civilian males or non-pregnant, non-lactating females
* Age 18-45
* Give informed consent and understand risk and benefit of study
* Understands and willing to comply with all protocol procedures and time commitment
* FEMALES only: surgically sterilized or received a negative pregnancy test on day of first injection AND agrees to practice adequate birth control, if necessary, for the next 7 months after first vaccination.

Exclusion Criteria:

* Currently has or has had a history of significant organ/system disease
* History of allergy to any vaccine
* Allergy to component of vaccine such as aluminum hydroxide
* Presence of significant unexplained laboratory abnormality
* HIV sero-positive or any other immunosuppressive state
* Positive test for HBsAg, or hepatitis C
* Ongoing drug abuse/dependence
* Received any live vaccine, experimental products or immunosuppressive therapy in the last 28 days or inactivated vaccine in the past 14 days, or received parenteral immunoglobulin or blood products within the past 3 months
* Intention to leave study area for an extended period of time during the study
* Females: positive urine pregnancy test prior to vaccination

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2005-12-05 (Actual); Primary Completion 2006-11-30 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barnett Gibbs, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR); Paul B Keiser, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Clinical Trials Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
WRAIR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 subjects were enrolled to be randomized into 1 of 3 cohorts at the WRAIR CTC.
Period: Overall Study
Arm/Group | 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant | 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D With Adjuvant | 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant
Started | 12 | 11 | 11
Completed | 9 | 8 | 9
Not Completed | 3 | 3 | 2
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant | 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D With Adjuvant | 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant | Total
Number analyzed (Participants) | 12 | 11 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.6 (9.3) | 33.4 (7.6) | 29.9 (8.4) | 31.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 17
  Male | 6 | 5 | 6 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — There is discrepancy in the demographic data within the Final Clinical Study Report (FCSR). Number of subject for 1) 25ug states total number of 12 subjects analyzed, but the race data indicates 13 subjects. Number of subjects for 2) 25ug states total number of 11 subjects analyzed, but the race data indicates 12 subjects analyzed. Data must me entered as indicated in the FCSR.
  Participants
    White | 7 | 5 | 4 | 16
    Black or African American | 5 | 7 | 7 | 19
    Hispanic or Latino | 1 | 1 | 1 | 3
    Asian | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Safety: Severity Summary of Solicited and Unsolicited Adverse Events
Description: Solicited and unsolicited summary of severity of adverse events (AEs) during the 7 day follow-up period after each vaccination
Time Frame: 7 day f/u period after each vaccination
Measure: Number; unit: AEs
Arm/Group | 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant | 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D With Adjuvant | 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant
Number analyzed (Participants) | 12 | 11 | 11
AEs
  Solicited: Mild | 67 | 92 | 70
  Solicited: Moderate | 3 | 16 | 10
  Solicited: Not related to study drug | 8 | 3 | 6
  Solicited: Related to study drug | 62 | 105 | 74
  Unsolicited: Number of subjects with atleast 1 AE | 10 | 10 | 7
  Unsolicited: Mild | 36 | 19 | 14
  Unsolicited: Moderate | 7 | 2 | 5
  Unsolicited: Severe | 4 | 2 | 2
  Unsolicited: Not related to study drug | 42 | 21 | 21
  Unsolicited: Related to study drug | 5 | 2 | 0

2. Primary Outcome: Safety: Adverse Event Type Summarized by Dose
Description: Adverse events summarized by type and dose
Time Frame: 7 days after each vaccination
Population: Both 25ug groups (1 and 2) were grouped for this analysis as both groups received the same dosage
Measure: Number; unit: Number of AEs
Groups:
- 25ug Group B Meningococcal 44/76 MOS NOMV 5D: Subjects received 25ug Group B Meningococcal 44/76 MOS NOMV 5D with and without AI (OH)3 adjuvant intramuscularly at 0, 6, and 24 weeks.
  25ug Group B Meningococcal 44/76 MOS NOMV 5D Vaccine: The study was conducted as a phase 1, outpatient, dose-escalating study for the Meningococcal 44/76 MOS NOMV 5D Vaccine (lot number 1119). 25µg with and without adjuvant were administered. Vaccinations were given intramuscularly at 0, 6, and 24 weeks.
- 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant: Subjects received 50ug Group B Meningococcal 44/76 MOS NOMV 5D without AI (OH)3 adjuvant intramuscularly at 0, 6, and 24 weeks.
  50ug Group B Meningococcal 44/76 MOS NOMV 5D Vaccine: The study was conducted as a phase 1, outpatient, dose-escalating study for the Meningococcal 44/76 MOS NOMV 5D Vaccine (lot number 1119). 50µg without adjuvant was administered. Vaccinations were given intramuscularly at 0, 6, and 24 weeks.
Arm/Group | 25ug Group B Meningococcal 44/76 MOS NOMV 5D | 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant
Number analyzed (Participants) | 23 | 11
Number of AEs
  Blood and lymphatic system disorders | 2 | 0
  Gastrointestinal disorders | 3 | 0
  General disorders | 65 | 75
  Infection and infestations | 5 | 7
  Injury, poisoning and procedural complications | 4 | 0
  Investigations | 8 | 1
  Metabolism and nutrition disorders | 2 | 0
  Musculoskeletal and connective tissue disorders | 8 | 8
  Nervous system disorders | 11 | 10
  Renal and urinary disorders | 5 | 0
  Respiratory, thoracic and mediastinal disorders | 3 | 0
  Skin and subcutaneous tissue disorders | 1 | 0

3. Secondary Outcome: Weeks to Serconversion
Description: Weeks to seroconversion evaluated by serum bactericidal assay. Immunogenicity was determined by assessing the number of subjects, in each cohort, who seroconverted. Seroconversion was defined as a 4-fold or greater increase in serum bactericidal antibodies against the vaccine strain. The geometric mean bactericidal titer (GMT) for each group was determined prior to vaccination and at 2 weeks after each vaccination. For each group, the GMT ratio relative to baseline and after 1, 2, or 3 vaccinations and the 95% 2-sided confidence interval was determined. A seroconversion of ≥50% of the subjects after 2 or more doses would meet the criteria for further vaccine development.
Time Frame: 26 weeks
Population: Number analyzed are subjects that seroconverted
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant | 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D With Adjuvant | 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant
Number analyzed (Participants) | 9 | 12 | 13
Weeks
  Test Antigen: 44/76: number analyzed (Participants) | 6 | 5 | 6
  Test Antigen: 44/76 | 2.0 (0.0) | 4.0 (4.5) | 3.0 (2.4)
  Test Antigen: 8570: number analyzed (Participants) | 1 | 1 | 2
  Test Antigen: 8570 | 8.0 (0.0) | 8.0 (0.0) | 8.0 (0.0)
  Test Antigen: 9162: number analyzed (Participants) | 1 | 2 | 2
  Test Antigen: 9162 | 26.0 (0.0) | 8.0 (0.0) | 8.0 (0.0)
  Test Antigen: 44/76 P: number analyzed (Participants) | 1 | 4 | 3
  Test Antigen: 44/76 P | 8.0 (0.0) | 12.5 (9.0) | 8.0 (0.0)

4. Secondary Outcome: Percentage of Subjects With 2-fold and 4-fold Increase IgG Antibody Conversion
Description: Percentage of subjects with ELISA 2-fold and 4-fold increase from baseline IgG antibody Conversion
Time Frame: 26 weeks
Population: Number of participants analyzed represents subjects who experienced increases from baseline
Measure: Number; unit: % of subjects
Arm/Group | 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant | 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D With Adjuvant | 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant
Number analyzed (Participants) | 10 | 9 | 10
% of subjects
  2-fold increase from BL: 44/76 NOMV IgG | 80.0 | 88.9 | 100.0
  2-fold increase from BL: L3, 7 LOS | 30.0 | 66.7 | 60.0
  2-fold increase from BL: GNA1870 | 0.0 | 66.7 | 50.0
  2-fold increase from BL: Opc | 60.0 | 33.3 | 80.0
  2-fold increase from BL: 44/76 P | 60.0 | 77.8 | 80.0
  4-fold increase from BL: 44/76 NOMV IgG | 20.0 | 55.6 | 70.0
  4-fold increase from BL: L3, 7 LOS | 10.0 | 22.2 | 10.0
  4-fold increase from BL: GNA1870 | 0.0 | 11.1 | 10.0
  4-fold increase from BL: Opc | 20.0 | 22.2 | 20.0
  4-fold increase from BL: 44/76 P | 40.0 | 22.2 | 50.0

ADVERSE EVENTS:
Time Frame: 7 days after each vaccination
Arm/Group | 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant | 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D With Adjuvant | 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1) 25ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant (N=12) | 2) 25ug Group B Meningococcal 44/76 MOS NOMV 5D With Adjuvant (N=11) | 3) 50ug Group B Meningococcal 44/76 MOS NOMV 5D w/o Adjuvant (N=11)
Pain (General disorders) | 12 (22) | 11 (52) | 11 (31)
Swelling (General disorders) | 5 (5) | 8 (8) | 7 (7)
Tenderness (Injury, poisoning and procedural complications) | 12 (17) | 11 (28) | 11 (21)
Pain lifting arm (General disorders) | 8 (8) | 11 (17) | 11 (13)
Warmth (General disorders) | 0 (0) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 9 (9) | 5 (5)
Induration (General disorders) | 2 (2) | 1 (1) | 1 (1)
Bruise (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypochromasia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin inconjugated increated (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Haptoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 6 (6)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No